CLINICAL TRIAL: NCT03113942
Title: Study of Pomalidomide in Anal Cancer Precursors (SPACE): a Phase 2 Study of Immunomodulation in People With Persistent HPV-associated High Grade Squamous Intraepithelial Lesions
Brief Title: Study of Pomalidomide in Anal Cancer Precursors
Acronym: SPACE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPACE
Record Dates: First submitted 2017-03-08; First posted 2017-04-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: High Grade Squamous Intra-epithelial Lesion (HSIL)
MeSH Terms: interventions — pomalidomide

STUDY DESIGN:
Intervention Model Description: Open label, phase 2 trial, single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pomalidomide group (Experimental): Open label - all participants will receive pomalidomide 2mg orally once a day for 6 cycles (21 days on treatment and a 7 day rest period constitutes a cycle).
  Interventions: Drug: Pomalidomide 2 MG Oral Capsule [Pomalyst]

INTERVENTIONS:
Drug: Pomalidomide 2 MG Oral Capsule [Pomalyst] — Pomalidomide is an oral immunomodulatory derivative of thalidomide. Thalidomide and its derivatives are small molecules with broad effects on immune activation, including T-cell activation and responsiveness. Pomalidomide augments T cell responsiveness and proliferation by several mechanisms, many mediated by transcriptional regulation downstream of its primary target, cereblon. Effects include increased production of IL-2 and interferon-γ (IFN-γ), enhanced CD4+ and CD8+ T cell co-stimulation.
  Other Names: pomalidomide; Pomalyst

SUMMARY:
This is a single centre open label phase II trial to determine the antitumor efficacy of the oral immunomodulatory agent pomalidomide in persistent human papillomavirus (HPV) -associated high grade squamous intra-epithelial lesions (HSIL) in patients with and without human immunodeficiency virus (HIV) infection.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent high grade squamous intra-epithelial lesion (HSIL) which must meet all of the following criteria:

   i. Pathologically confirmed grade 2 or 3 AIN demonstrated by high resolution anoscopy with grade on each occasion re-confirmed at screening by nominated study pathologist from Douglas Hanly Moir (DHM) (pathology case review to be conducted prior to enrolment) ii. Lesion must have been visualised on at least three sequential occasions over at least 12 months, including the pre enrolment screening high resolution anoscopy (HRA).

   iii. Lesion must have persistent geographical characteristics consistent with a single lesion observed over time (as defined in the Manual of Operations).
2. No history of thromboembolic disease
3. No evidence of anal cancer or Superficially Invasive Squamous Cell Carcinoma of the Anus (SISCCA)
4. Willingness to use appropriate contraception (including refraining from sperm donation)
5. Age 18 years or older
6. Provision of written informed consent

   In addition, for subjects with HIV:
7. Adherence to a stable suppressive antiretroviral therapy (ART) regimen, unchanged for at least two months
8. CD4+ count ≥ 200 cells/µl
9. HIV viral load < 200 copies/mL for at least six months

Exclusion Criteria:

1. Absolute neutrophil count (ANC) <1000 cells/μL
2. Haemoglobin <10.0 g/dL
3. Platelet count <75,000 cells/μL
4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > three times upper limit of normal
5. Calculated or measured creatinine clearance (CLCr) ≤ 50 mL/min (calculated by Cockcroft-Gault formula)
6. Patients with significant cardiac dysfunction including congestive heart failure, NY Heart Association Class II; Myocardial infarction within 12 months of starting study; unstable of poorly controlled angina
7. Current pregnancy or breastfeeding
8. Any condition not already outlined above which, in the opinion of the clinical investigator, would place the subject at risk if they participated or would jeopardise adherence or follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Histological High Grade Squamous Intraepithelial Lesions (HSIL) clearance at 6 months of therapy | 6 months
  Histological high grade squamous intra-epithelial lesion clearance

SECONDARY OUTCOMES:
incidence of grade 3 and 4 adverse events and therapy delays (tolerability) | 6 months
  incidence of grade 3 and 4 adverse events and therapy delays (tolerability)
number of subjects completing of full six month course | 6 months
  number of subjects completing of full six month course (feasibility of polidamide in this setting)
effect of pomalidomide on self-reported health related quality of life and cancer anxiety during and after therapy | 6 months
  individual patient change in quality of life questionnaire (SF12) from baseline to mid therapy and end therapy

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's Hospital, Darlinghurst, New South Wales, Australia

REFERENCES:
- [Background] Munoz N, Castellsague X, Berrington de Gonzalez A, Gissmann L. Chapter 1: HPV in the etiology of human cancer. Vaccine. 2006 Aug 31;24 Suppl 3:S3/1-10. doi: 10.1016/j.vaccine.2006.05.115. Epub 2006 Jun 23. PMID 16949995
- [Background] Parkin DM, Bray F. Chapter 2: The burden of HPV-related cancers. Vaccine. 2006 Aug 31;24 Suppl 3:S3/11-25. doi: 10.1016/j.vaccine.2006.05.111. PMID 16949997
- [Background] World Health Organization International Agency for Reseach on Cancer. IARC Monograph on the Evaluation of Carcinogenic Risks to Humans: Volume 90, Human Papillomavirus. World Health Organization, Geneva 2007.
- [Background] Machalek DA, Poynten M, Jin F, Fairley CK, Farnsworth A, Garland SM, Hillman RJ, Petoumenos K, Roberts J, Tabrizi SN, Templeton DJ, Grulich AE. Anal human papillomavirus infection and associated neoplastic lesions in men who have sex with men: a systematic review and meta-analysis. Lancet Oncol. 2012 May;13(5):487-500. doi: 10.1016/S1470-2045(12)70080-3. Epub 2012 Mar 23. PMID 22445259
- [Background] Palefsky JM. Anal cancer prevention in HIV-positive men and women. Curr Opin Oncol. 2009 Sep;21(5):433-8. doi: 10.1097/CCO.0b013e32832f511a. PMID 19587592
- [Background] Grulich AE, Poynten IM, Machalek DA, Jin F, Templeton DJ, Hillman RJ. The epidemiology of anal cancer. Sex Health. 2012 Dec;9(6):504-8. doi: 10.1071/SH12070. PMID 22958581
- [Background] Petoumenos K, van Leuwen MT, Vajdic CM, Woolley I, Chuah J, Templeton DJ, Grulich AE, Law MG; Australian HIV Observational Database. Cancer, immunodeficiency and antiretroviral treatment: results from the Australian HIV Observational Database (AHOD). HIV Med. 2013 Feb;14(2):77-84. doi: 10.1111/j.1468-1293.2012.01038.x. Epub 2012 Aug 30. PMID 22934689
- [Background] Yarchoan R, Tosato G, Little RF. Therapy insight: AIDS-related malignancies--the influence of antiviral therapy on pathogenesis and management. Nat Clin Pract Oncol. 2005 Aug;2(8):406-15; quiz 423. doi: 10.1038/ncponc0253. PMID 16130937
- [Background] Ajani JA, Winter KA, Gunderson LL, Pedersen J, Benson AB 3rd, Thomas CR Jr, Mayer RJ, Haddock MG, Rich TA, Willett C. Fluorouracil, mitomycin, and radiotherapy vs fluorouracil, cisplatin, and radiotherapy for carcinoma of the anal canal: a randomized controlled trial. JAMA. 2008 Apr 23;299(16):1914-21. doi: 10.1001/jama.299.16.1914. PMID 18430910
- [Background] Moscicki AB, Schiffman M, Kjaer S, Villa LL. Chapter 5: Updating the natural history of HPV and anogenital cancer. Vaccine. 2006 Aug 31;24 Suppl 3:S3/42-51. doi: 10.1016/j.vaccine.2006.06.018. Epub 2006 Jun 23. PMID 16950017
- [Background] Tong WW, Shepherd K, Garland S, Meagher A, Templeton DJ, Fairley CK, Jin F, Poynten IM, Zaunders J, Hillman RJ, Grulich AE, Kelleher AD, Carr A; Study of the Prevention of Anal Cancer (SPANC) team. Human papillomavirus 16-specific T-cell responses and spontaneous regression of anal high-grade squamous intraepithelial lesions. J Infect Dis. 2015 Feb 1;211(3):405-15. doi: 10.1093/infdis/jiu461. Epub 2014 Aug 19. PMID 25139018
- [Background] Quach H, Ritchie D, Stewart AK, Neeson P, Harrison S, Smyth MJ, Prince HM. Mechanism of action of immunomodulatory drugs (IMiDS) in multiple myeloma. Leukemia. 2010 Jan;24(1):22-32. doi: 10.1038/leu.2009.236. Epub 2009 Nov 12. PMID 19907437
- [Background] Ito T, Ando H, Suzuki T, Ogura T, Hotta K, Imamura Y, Yamaguchi Y, Handa H. Identification of a primary target of thalidomide teratogenicity. Science. 2010 Mar 12;327(5971):1345-50. doi: 10.1126/science.1177319. PMID 20223979
- [Background] Gorgun G, Calabrese E, Soydan E, Hideshima T, Perrone G, Bandi M, Cirstea D, Santo L, Hu Y, Tai YT, Nahar S, Mimura N, Fabre C, Raje N, Munshi N, Richardson P, Anderson KC. Immunomodulatory effects of lenalidomide and pomalidomide on interaction of tumor and bone marrow accessory cells in multiple myeloma. Blood. 2010 Oct 28;116(17):3227-37. doi: 10.1182/blood-2010-04-279893. Epub 2010 Jul 22. PMID 20651070
- [Background] Lentzsch S, LeBlanc R, Podar K, Davies F, Lin B, Hideshima T, Catley L, Stirling DI, Anderson KC. Immunomodulatory analogs of thalidomide inhibit growth of Hs Sultan cells and angiogenesis in vivo. Leukemia. 2003 Jan;17(1):41-4. doi: 10.1038/sj.leu.2402745. PMID 12529658
- [Background] Reddy N, Hernandez-Ilizaliturri FJ, Deeb G, Roth M, Vaughn M, Knight J, Wallace P, Czuczman MS. Immunomodulatory drugs stimulate natural killer-cell function, alter cytokine production by dendritic cells, and inhibit angiogenesis enhancing the anti-tumour activity of rituximab in vivo. Br J Haematol. 2008 Jan;140(1):36-45. doi: 10.1111/j.1365-2141.2007.06841.x. Epub 2007 Nov 9. PMID 17995965
- [Background] Verhelle D, Corral LG, Wong K, Mueller JH, Moutouh-de Parseval L, Jensen-Pergakes K, Schafer PH, Chen R, Glezer E, Ferguson GD, Lopez-Girona A, Muller GW, Brady HA, Chan KW. Lenalidomide and CC-4047 inhibit the proliferation of malignant B cells while expanding normal CD34+ progenitor cells. Cancer Res. 2007 Jan 15;67(2):746-55. doi: 10.1158/0008-5472.CAN-06-2317. PMID 17234786
- [Background] Zhu D, Corral LG, Fleming YW, Stein B. Immunomodulatory drugs Revlimid (lenalidomide) and CC-4047 induce apoptosis of both hematological and solid tumor cells through NK cell activation. Cancer Immunol Immunother. 2008 Dec;57(12):1849-59. doi: 10.1007/s00262-008-0512-7. Epub 2008 Apr 8. PMID 18392823
- [Background] Shalapour S, Zelmer A, Pfau M, Moderegger E, Costa-Blechschmidt C, van Landeghem FK, Taube T, Fichtner I, Buhrer C, Henze G, Seeger K, Wellmann S. The thalidomide analogue, CC-4047, induces apoptosis signaling and growth arrest in childhood acute lymphoblastic leukemia cells in vitro and in vivo. Clin Cancer Res. 2006 Sep 15;12(18):5526-32. doi: 10.1158/1078-0432.CCR-06-0719. PMID 17000689
- [Background] Escoubet-Lozach L, Lin IL, Jensen-Pergakes K, Brady HA, Gandhi AK, Schafer PH, Muller GW, Worland PJ, Chan KW, Verhelle D. Pomalidomide and lenalidomide induce p21 WAF-1 expression in both lymphoma and multiple myeloma through a LSD1-mediated epigenetic mechanism. Cancer Res. 2009 Sep 15;69(18):7347-56. doi: 10.1158/0008-5472.CAN-08-4898. Epub 2009 Sep 8. PMID 19738071
- [Background] Pal R, Monaghan SA, Hassett AC, Mapara MY, Schafer P, Roodman GD, Ragni MV, Moscinski L, List A, Lentzsch S. Immunomodulatory derivatives induce PU.1 down-regulation, myeloid maturation arrest, and neutropenia. Blood. 2010 Jan 21;115(3):605-14. doi: 10.1182/blood-2009-05-221077. Epub 2009 Nov 25. PMID 19965623
- [Background] Polizzotto MN, Sereti I, Uldrick TS, et al. Pomalidomide induces expansion of activated and central memory CD4 and CD8 T-cells in vivo in patients with and without HIV infection. American Society of Hematology Annual Meeting, San Francisco 2014.
- [Background] Polizzotto MN, Uldrick TS, Wyvill KM, Aleman K, Peer CJ, Bevans M, Sereti I, Maldarelli F, Whitby D, Marshall V, Goncalves PH, Khetani V, Figg WD, Steinberg SM, Zeldis JB, Yarchoan R. Pomalidomide for Symptomatic Kaposi's Sarcoma in People With and Without HIV Infection: A Phase I/II Study. J Clin Oncol. 2016 Dec;34(34):4125-4131. doi: 10.1200/JCO.2016.69.3812. Epub 2016 Oct 31. PMID 27863194
- [Background] Machalek DA, Grulich AE, Hillman RJ, Jin F, Templeton DJ, Tabrizi SN, Garland SM, Prestage G, McCaffery K, Howard K, Tong W, Fairley CK, Roberts J, Farnsworth A, Poynten IM; SPANC Study Team. The Study of the Prevention of Anal Cancer (SPANC): design and methods of a three-year prospective cohort study. BMC Public Health. 2013 Oct 9;13:946. doi: 10.1186/1471-2458-13-946. PMID 24107134
- [Background] Richel O, de Vries HJ, van Noesel CJ, Dijkgraaf MG, Prins JM. Comparison of imiquimod, topical fluorouracil, and electrocautery for the treatment of anal intraepithelial neoplasia in HIV-positive men who have sex with men: an open-label, randomised controlled trial. Lancet Oncol. 2013 Apr;14(4):346-53. doi: 10.1016/S1470-2045(13)70067-6. Epub 2013 Mar 15. PMID 23499546
- [Background] POMALYST® (pomalidomide) capsules Product Information. Department of Health Therapeutic Goods Administration (TGA) April 2016. https://www.ebs.tga.gov.au/ebs/picmi/picmirepository.nsf/pdf accessed 23 Nov 2016.